CLINICAL TRIAL: NCT03154528
Title: Role of Vitamin D in Androgenetic Alopecia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Miral Hassan, principle investigator, Assiut University
Other Study IDs: MAGA2017
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Alopecia, Androgenetic
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control group: serum level of Vitamin D is going to be checked by ELISA in 30 healthy control volunteers
  Interventions: Diagnostic Test: serum vitamin D level by ELISA
- case study group: serum level of Vitamin D is going to be checked by ELISA in 60 Androgenetic Alopecia patients.
  Interventions: Diagnostic Test: serum vitamin D level by ELISA

INTERVENTIONS:
Diagnostic Test: serum vitamin D level by ELISA — The study will include 60 patients with androgenetic alopecia (30 males & 30 females) and 30 age and sex-matched healthy volunteers. Study subjects will be recruited from the Dermatology Outpatients' Clinic, Assiut University Hospitals, Assiut, Egypt. Informed consent will be obtained from all subjects

SUMMARY:
Androgenetic alopecia is a common form of diffuse hair loss in both men and women,It primarily affects the top and front of the scalp with different clinical presentations and there are numerous classification systems for grading purposes.

DETAILED DESCRIPTION:
These systems vary from the simple systems based on recession of the hairline to more advanced multifactorial systems based on morphological and dynamic parameters that affect the scalp and hair. Most of these systems have certain limitations. Currently, the most commonly used are Hamilton- Norwood classification system for males where there are two areas of hair loss that gradually enlarge to produce recession at the temples and thinning in the crown. These regions coalesce until the entire front, top and crown (vertex) of the scalp are bald(2 major pattern,7 grades) and the Ludwig system for females which classify the Female Pattern Hair Loss into three grades depending on the reduction in hair density over the crown and frontal scalp with retention of the frontal hairline.

Etiopathogenesis of Androgenetic Alopecia has not yet been fully elucidated. Genetic factors, hair follicle cycle abnormalities, aging process and androgen dependent process including end organ sensitivity have been all incriminated as etiological factors .

Dermoscopy has emerged as an useful tool in the diagnosis of hair loss disorder including Androgenetic Alopecia. Important features of Androgenetic Alopecia on Dermoscopy include hair shaft thickness heterogeneity, yellow dots (irregularly distributed and with a remarkable variability in size and shape), perifollicular discolouration (the peripilar sign), an increased proportion of thin and vellus hairs (>10 % of the hairs) and a large number of follicular units with only one emerging hair shaft. Thin wavy hair and honeycomb hyperpigmentation often coexist as additional, nonspecific features Vitamin D is a secosteroid hormone that plays an important role in calcium homeostasis and bone health. It has three sources: endogenous synthesis in the skin, which is induced by Ultraviolet B radiation; dietary intake; and supplementation .

Basically, Vitamin D is a modulator of both innate and adaptive immune systems through its various effects on T and B lymphocytes, dendritic cells and macrophages. There is a well-established causal connection between vitamin D deficiency and some autoimmune diseases , and possible association with some hair disorders, as it has been demonstrated that vitamin D receptors are strongly expressed in hair follicles and keratinocytes. Such an expression was found to be necessary for maintenance of the normal hair cycle. Also, it has also been shown that lack of vitamin D receptors reduces epidermal differentiation and hair follicle growth, and that an optimum concentration of Vitamin D3 is essential to delay aging and hair loss.

Several studies were done to evaluate the role of vitamin D in different hair disorders with contrasting results. Some studies revealed low serum levels of Vitamin D in women with chronic telogen effluvium,Female Pattern Hair Loss and Alopecia Areata.While, two studies showed no correlation between the extent and severity of male androgenetic alopecia with serum Vitamin D3 level.

Based on the above contrasting reports, we sought to evaluate the levels of Vitamin D in patients with androgenetic alopecia in order to establish its possible role in the etiopathogenesis and hence in the treatment of such a common and chronic hair disorder

ELIGIBILITY:
Inclusion Criteria:

* The study will include 60 patients with androgenetic alopecia (30 males & 30 females) and 30 age and sex-matched healthy volunteers.

Exclusion Criteria:

- 1-Patients with a history of topical or systemic treatment within the last month.

2-Patients with a history of concomitant skin or systemic disease. 3- Pregnant or lactating women. 4- Smokers. 5- Patients receiving phototherapy within 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include 60 patients with androgenetic alopecia (30 males & 30 females) and 30 age and sex-matched healthy volunteers. Study subjects will be recruited from the Dermatology Outpatients' Clinic, Assiut University Hospitals, Assiut, Egypt. Informed consent will be obtained from all subjects
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-03-30 (Estimated); Primary Completion 2019-08-21 (Estimated); Study Completion 2019-12-12 (Estimated)

PRIMARY OUTCOMES:
Serum Vitamin D level | 1 year
  Laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Miral Taya, MD, Principal Investigator — Assiut Uneversity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varothai S, Bergfeld WF. Androgenetic alopecia: an evidence-based treatment update. Am J Clin Dermatol. 2014 Jul;15(3):217-30. doi: 10.1007/s40257-014-0077-5. PMID 24848508
- [Result] Gupta M, Mysore V. Classifications of Patterned Hair Loss: A Review. J Cutan Aesthet Surg. 2016 Jan-Mar;9(1):3-12. doi: 10.4103/0974-2077.178536. PMID 27081243
- [Result] Vujovic A, Del Marmol V. The female pattern hair loss: review of etiopathogenesis and diagnosis. Biomed Res Int. 2014;2014:767628. doi: 10.1155/2014/767628. Epub 2014 Apr 9. PMID 24812631
- [Result] Orme S, Cullen DR, Messenger AG. Diffuse female hair loss: are androgens necessary? Br J Dermatol. 1999 Sep;141(3):521-3. doi: 10.1046/j.1365-2133.1999.03049.x. PMID 10583059
- [Result] Kaliyadan F, Nambiar A, Vijayaraghavan S. Androgenetic alopecia: an update. Indian J Dermatol Venereol Leprol. 2013 Sep-Oct;79(5):613-25. doi: 10.4103/0378-6323.116730. PMID 23974579
- [Result] Errichetti E, Stinco G. Dermoscopy in General Dermatology: A Practical Overview. Dermatol Ther (Heidelb). 2016 Dec;6(4):471-507. doi: 10.1007/s13555-016-0141-6. Epub 2016 Sep 9. PMID 27613297
- [Result] Bikle DD. Vitamin D metabolism and function in the skin. Mol Cell Endocrinol. 2011 Dec 5;347(1-2):80-9. doi: 10.1016/j.mce.2011.05.017. Epub 2011 Jun 1. PMID 21664236
- [Result] Arnson Y, Amital H, Shoenfeld Y. Vitamin D and autoimmunity: new aetiological and therapeutic considerations. Ann Rheum Dis. 2007 Sep;66(9):1137-42. doi: 10.1136/ard.2007.069831. Epub 2007 Jun 8. PMID 17557889
- [Result] Malloy PJ, Feldman D. The role of vitamin D receptor mutations in the development of alopecia. Mol Cell Endocrinol. 2011 Dec 5;347(1-2):90-6. doi: 10.1016/j.mce.2011.05.045. Epub 2011 Jun 13. PMID 21693169
- [Result] Amor KT, Rashid RM, Mirmirani P. Does D matter? The role of vitamin D in hair disorders and hair follicle cycling. Dermatol Online J. 2010 Feb 15;16(2):3. PMID 20178699
- [Result] Rasheed H, Mahgoub D, Hegazy R, El-Komy M, Abdel Hay R, Hamid MA, Hamdy E. Serum ferritin and vitamin d in female hair loss: do they play a role? Skin Pharmacol Physiol. 2013;26(2):101-7. doi: 10.1159/000346698. Epub 2013 Feb 20. PMID 23428658
- [Result] Banihashemi M, Nahidi Y, Meibodi NT, Jarahi L, Dolatkhah M. Serum Vitamin D3 Level in Patients with Female Pattern Hair Loss. Int J Trichology. 2016 Jul-Sep;8(3):116-20. doi: 10.4103/0974-7753.188965. PMID 27625563
- [Result] Bakry OA, El Farargy SM, El Shafiee MK, Soliman A. Serum Vitamin D in patients with alopecia areata. Indian Dermatol Online J. 2016 Sep-Oct;7(5):371-377. doi: 10.4103/2229-5178.190504. PMID 27730032
- [Result] Bolland MJ, Ames RW, Grey AB, Horne AM, Mason BH, Gamble GD, Reid IR. Does degree of baldness influence vitamin D status? Med J Aust. 2008 Dec 1-15;189(11-12):674-5. doi: 10.5694/j.1326-5377.2008.tb02241.x. PMID 19061473